CLINICAL TRIAL: NCT06951828
Title: A Phase I, Randomized, Open-label, Two-Arm, Parallel Group, Single-Dose Study to Compare the Pharmacokinetics, Safety and Immunogenicity of the Auto-injector and Pre-filled Syringe of CT-P43 in Healthy Male Subjects
Brief Title: A Study to Compare the Auto-injector and Pre-filled Syringe of CT-P43 in Healthy Male Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CT-P43 1.3
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CT-P43 Auto-injector (Experimental): CT-P43, 45 mg in 0.5 ml, a single subcutaneous (SC) injection via auto-injector (AI)
  Interventions: Biological: CT-P43
- CT-P43 Pre-filled syringe (Active Comparator): CT-P43, 45 mg in 0.5 ml, a single SC injection via pre-filled syringe (PFS)
  Interventions: Biological: CT-P43

INTERVENTIONS:
Biological: CT-P43 — CT-P43, 45 mg in 0.5 ml, a single subcutaneous (SC) injection via auto-injector (AI)
  Arms: CT-P43 Auto-injector
Biological: CT-P43 — CT-P43, 45 mg in 0.5 ml, a single subcutaneous (SC) injection via pre-filled syringe (PFS)
  Arms: CT-P43 Pre-filled syringe

SUMMARY:
This is phase 1 study to Compare the Pharmacokinetics, Safety and Immunogenicity of the Auto-injector and Pre-filled syringe of CT-P43 in Healthy Male Subjects.

DETAILED DESCRIPTION:
CT-P43, containing the active ingredient ustekinumab, is being developed by CELLTRION, Inc. as a proposed biosimilar to the reference product, Stelara. In this study, Pharmacokinetics, Safety and Immunogenicity of the Auto-injector and Pre-filled syringe of CT-P43 will be evaluated in Healthy Male Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, between the ages of 19 and 55 years, both inclusive.
* Subject has a body weight between 60 to 90 kg, both inclusive, and a BMI between 18.5 and 29.9 kg/m2, both inclusive, when rounded to the nearest tenth.

Exclusion Criteria:

* A medical history and/or condition that is considered significant
* Clinically significant allergic reactions, hypersensitivity
* History or current infection of hepatitis B virus, hepatitis C virus, human immunodeficiency virus, or syphilis
* Active or latent Tuberculosis
* History of malignancy
* Previous exposure to ustekinumab or a biosimilar of ustekinumab or any drug that directly targets interleukin (IL)-12, IL-17 or IL-23

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
PK similarity demonstration by AUC 0-inf | Day113
  Demonstrate the PK similarity in terms of area under the concentration-time curve from time zero to infinity (AUC0-inf) of CT-P43 SC administration via AI versus PFS in healthy male subjects up to Day 113 (Week 16).
PK similarity demonstration by Cmax | Day113
  Demonstrate the PK similarity in terms of maximum serum concentration (Cmax) of CT-P43 SC administration via AI versus PFS in healthy male subjects up to Day 113 (Week 16).

SECONDARY OUTCOMES:
Additional PK evaluation | Day113
  Evaluate additional PK in terms of AUC from time zero to the last quantifiable concentration (AUC0-last). Time to maximum concentration (Tmax), Terminal half-life (t1/2), Percentage of AUC0-inf obtained by extrapolation (%AUCextrap).
Safety evaluation by AEs | Day113
  Evaluate safety in terms of adverse events (including treatment-emergent adverse events [TEAEs] and serious adverse events[SAEs]).

CONTACTS AND LOCATIONS:
Overall Officials: Hyewon Chung, Principal Investigator — Korea University Guro Hospital (Department of Clinical Pharmacology)
Locations (1):
- Korea University Guro Hospital, Seoul, Guro-gu, South Korea